30.04.2019

## Eskisehir Osmangazi University Department of Algology Eskisehir/Turkey

Comparison of the effect of ultrasound-guided greater occipital nerve block and pulsed radiofrequency therapy in patients with chronic migraine

Informed Consent Form

In the study, Comparison of the effect of ultrasound-guided greater occipital nerve block and pulsed radiofrequency therapy in patients with chronic migraine, to be carried out at Eskişehir Osmangazi University, two treatment options to be applied randomly are used to reduce the number and severity of attacks in chronic migraine patients. As a result of these treatments, there is no reduction in pain, minor bleeding in the area, and there is a risk of infection if the rules of asepsis are not followed.

The risks and expected benefits of both treatment methods were explained to me. I was told to apply to the clinic, which I can always reach and access in unexpected situations.(Contact number: 0222 239 29 79)

I willingly and voluntarily agree to participate in the study Comparison of the effectiveness of ultrasound-guided greater occipital nerve block and pulsed radiofrequency therapy in patients with chronic migraine.

| Patient name and surname: |
|---------------------------|
| Patient protocol: |
| Date: |
| Patient signature: |